CLINICAL TRIAL: NCT04793607
Title: Interventions for Malignant Pleural Effusions Impact on Fatigue Study
Brief Title: Interventions for Malignant Pleural Effusions Impact on Fatigue
Acronym: IMPE-F
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Collaborators: Rocket Medical plc (Other)
Responsible Party: Sponsor
Other Study IDs: NHCT0161
Record Dates: First submitted 2020-08-13; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Malignant Pleural Effusion
Keywords: pleural effusion; malignancy
MeSH Terms: conditions — Pleural Effusion, Malignant; Pleural Effusion; Neoplasms | interventions — Thoracoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pleural procedures — Any pleural procedure that removes fluid

SUMMARY:
Malignant Pleural Effusions (MPE) are a common problem with around 40,000 new cases in the UK each year. The presence of an MPE suggests a poor prognosis of on average of 3-12 months. It is therefore vital that the investigators consider how respiratory and palliative care physicians can best support patients with MPEs to have the best quality of life possible.

Breathlessness is the most common presenting symptom of an MPE and so impact on this has previously been studied . Cancer-related fatigue is very common with evidence suggesting around 40% of patients experience fatigue at diagnosis and up to 90% during anti-cancer treatment such as radiotherapy or chemotherapy. Review of the literature suggests that whether interventions to manage MPEs can improve patient fatigue has not previously been studied.

The aim of this study is to assess if interventions for MPEs could potentially improve patient fatigue as this information will be valuable for both patients and referring health-care professionals when making the decision of whether to have a procedure or not and build on the current evidence base around management of MPEs.

The study will be part of a Masters in Clinical Research and will be within a single trust. It will be a pilot study for a potentially larger multi-center study. With this in mind, aspects of how the study runs and notes on how it could be improved upon will be carefully recorded.

DETAILED DESCRIPTION:
The aim of the study is to assess if the interventions for MPEs have an impact on fatigue levels. There are multiple different possible interventions to treat a pleural effusion and the most appropriate is decided on a case-by-case basis after discussion between the patient and doctor. The study will have no impact on which intervention the participant receives.

Fatigue is extreme tiredness unrelieved by rest. It is how the patient feels and so there is no specific test for it. However there are a number of tools that help record a patients self-reported fatigue levels and how this changes over time. The FACIT-fatigue tool has been studied in patients with cancer-related fatigue and has the strongest evidence base and validation in this patient group. It involves the patient answering 13 questions related to fatigue and its impact on their activities of daily living.

There are multiple contributing factors associated with malignancy-related fatigue and so consent will be gained to gather data on potential confounding factors. This will include

* Patient age
* Sex
* Patient diagnosis (site/type of cancer and whether metastatic)
* Comorbidities (esp. lung disease)
* Time since cancer diagnosis
* Time since last anti-cancer therapy/if currently having chemotherapy or radiotherapy
* BEDS&GADS score for anxiety/depression
* Patient Outcome Score (POS) indicating whether high symptom burden
* Size of pleural effusion & if unilateral/bilateral
* Performance status
* Blood markers- Haemoglobin level & Creatinine

The study will involve a single pleural service in Northumbria Healthcare NHS Foundation Trust.

Both inpatients and outpatients are referred to the pleural service. They are assessed in clinic and a decision made on the most appropriate treatment of the Malignant Pleural Effusion. The study will have no impact on which intervention is chosen. Once the decision is made the patient will be asked by the doctor in clinic if they are potentially interested in being involved in the study. If they are interested then they will be seen by the researcher who will take them through the Participant Information Sheet (PIS) and give them the opportunity to ask questions. If they agree then they will be invited to provide written informed consent.

The researcher is a consultant with training in assessing patients capacity and so it will be ensured that all participants are able to give valid written consent. Those unable to give consent will be excluded from the study. Reasonable adjustments will be made to cater for patients with hearing or visual impairment.

It will be made clear that the decision to take part in the study or not will have no impact on the patient's care. It will also be explained that the patient is free to withdraw from the study at any time and under no obligation to give reason for doing so.

It will be made clear to the potential participants that taking part in the study will have no impact on their treatment. There will be no direct benefit to the participant other than for altruistic reasons such as knowing that their involvement is contributing to the research base which may improve care for patients of the future.

This study is fairly low burden as it is a short questionnaire about fatigue levels (13 questions) and permission to gather further data about the patient (age, sex, disease site, performance status, last Hb result- see list above). The participant will give permission for the researcher to telephone them to repeat the questions after 7,14 & 30 days. The question takes less than 5 minutes to answer and so is of low burden.

There is no direct risk to staff or patient.

It is possible that the patient becomes more unwell or dies during the 30-day study period. It may therefore be upsetting to the patient or family to be contacted if this was the case. To try and avoid this then the patient's electronic records will be consulted prior to making contact via telephone. However, it may occasionally be possible that the death is not yet recorded in the electronic records and so all calls will be handled in a sensitive manner. The researcher is a Palliative Medicine consultant with advanced communication skills training and many years experience of having discussions with patients approaching the end of life as well as bereaved families.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the Northumbria specialist pleural service to have an intervention for a malignant pleural effusion
* Age 18+ years

Exclusion Criteria:

° Patients who lack capacity to give consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient above the age of 18 with a presumed malignant pleural effusion referred to the Northumbria specialist pleural service
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue levels as measured by the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) form. Minimum score is zero and maximum score is 52. Higher scores mean high levels of fatigue. | Up to 1 month
  At the time of their pleural procedures, recruited participants will fill in, with the help of the investigator, the FACIT-F form to determine their current level of fatigue. The participant will then be contacted to record their fatigue levels using the same questionnaire at 7, 14 and 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Donna Wakefield, MBBS, Principal Investigator — Northumbria Healthcare NHS Foundation Trust
Locations (1):
- Northumbria HealthCare NHS Foundation Trust, Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feller-Kopman DJ, Reddy CB, DeCamp MM, Diekemper RL, Gould MK, Henry T, Iyer NP, Lee YCG, Lewis SZ, Maskell NA, Rahman NM, Sterman DH, Wahidi MM, Balekian AA. Management of Malignant Pleural Effusions. An Official ATS/STS/STR Clinical Practice Guideline. Am J Respir Crit Care Med. 2018 Oct 1;198(7):839-849. doi: 10.1164/rccm.201807-1415ST. PMID 30272503
- [Result] Hofman M, Ryan JL, Figueroa-Moseley CD, Jean-Pierre P, Morrow GR. Cancer-related fatigue: the scale of the problem. Oncologist. 2007;12 Suppl 1:4-10. doi: 10.1634/theoncologist.12-S1-4. PMID 17573451
- [Result] Minton O, Stone P. A systematic review of the scales used for the measurement of cancer-related fatigue (CRF). Ann Oncol. 2009 Jan;20(1):17-25. doi: 10.1093/annonc/mdn537. Epub 2008 Aug 4. PMID 18678767
- [Result] Prue G, Rankin J, Allen J, Gracey J, Cramp F. Cancer-related fatigue: A critical appraisal. Eur J Cancer. 2006 May;42(7):846-63. doi: 10.1016/j.ejca.2005.11.026. Epub 2006 Feb 7. PMID 16460928

DOCUMENTS (1):
  • Informed Consent Form (2020-07-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT04793607/ICF_000.pdf